CLINICAL TRIAL: NCT05222945
Title: ANRS EP69 BICTEVOIR : A Prospective Study to Determine the Cartography of Virologic Reservoir Related to Antiretroviral Concentrations in HIV-1 Chronic Patients Treated by a First Line Treatment Containing bictégravir, Emtricitabine and ténofovir alafénamide
Brief Title: A Study to Determine the Cartography of Virologic Reservoir Related to Antiretroviral Concentrations in HIV-1 Chronic Patients Treated by a First Line Treatment Containing bictégravir, Emtricitabine and ténofovir alafénamide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS EP69 BICTEVOIR
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: HIV-1-infection
Keywords: Viral cartography; Viral reservoir; Antiretroviral treatments diffusion
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm composed by 34 HIV-1 infected male subjects (Other)
  Interventions: Other: Biopsies and bloood samplings

INTERVENTIONS:
Other: Biopsies and bloood samplings — blood samples, rectal biopsies, nodes biopsies, cutaneous fat tissues biopsies, semen sample

SUMMARY:
The main objective of the study is to evaluate the diffusion of bictegravir and associated backbone (tenofovir alafenamide and emtricitabine) in HIV-1 chronic patients in the main putative reservoirs, namely inguinal lymph nodes, rectal, fat tissues and sperm.

DETAILED DESCRIPTION:
ANRS EP69 BICTEVOIR is an interventional pilot study, multicenter, involving the use of human biological samples.

34 HIV-1 infected male subjects, from Bicetre, La Pitié Salpêtriere, Antoine-Béclère, Necker, Hôtel-Dieu and Saint-Antoine Hospitals will be recruited.

Different samples will be performed during one single day:

* blood samples
* rectal biopsies
* nodes biopsies
* cutaneous fat tissues biopsies
* semen sample (at home)

ELIGIBILITY:
Inclusion Criteria:

* Male HIV-1 infected subjects
* Age > or = 18 years old
* Currently receiving as first line a stable ARV regimen containing bictegravir (at 50 mg once a day) and two nucleoside reverse transcriptase inhibitors, tenofovir alafenamide/emtricitabine (Biktarvy)
* HIV RNA <50 Cp/mL, undetectable 6 months after treatment initiation and confirmed and 12 months after treatment initiation.
* Normal laboratory value of TP and TCA and platelets numbers at screening
* Written and informed consent signed by the person and the investigator (no later than the day of pre-inclusion and prior to any examination realized in the frame of the research / study / trial) (article L1122-1-1 of the Public Health Code)
* Person affiliated or beneficiary of a social security scheme (article L1121-11 of the Public Health Code) (State Medical Aid or AME is not a social security scheme)

Exclusion Criteria:

* Single HIV-2 infection
* Biopsies contraindication, taking anticoagulant and antiplatelet drugs are not allowed
* Haemophilia
* Symptomatic sexually transmitted infection
* Being under guardianship or trusteeship mandate for future protection
* Participate to another research involving human person, categories 1 or 2,
* Associated treatments : carbamazepine, oxcarbazepine, phenytoin, phenobarbital, rifampicin, St. John's Wort.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of the diffusion of bictegravir and associated backbone (tenofovir alafenamide and emtricitabine) in sperm | At Day 0, At time T0 (before taking treatments)
  Dosage of the different antiretroviral drugs molecules in sperm
Characterization of the diffusion of bictegravir and associated backbone (tenofovir alafenamide and emtricitabine) in lymph nodes | At Day 0, between T1 (maximum 3 hours after tacking treatments) and T3 (8 hours after taking treatments)
  Dosage of the different antiretroviral drugs molecules in lymph nodes
Characterization of the diffusion of bictegravir and associated backbone (tenofovir alafenamide and emtricitabine) in fat tissues | At Day 0, between T1 (maximum 3 hours after tacking treatments) and T3 (8 hours after taking treatments)
  Dosage of the different antiretroviral drugs molecules in fat tissues
Characterization of the diffusion of bictegravir and associated backbone (tenofovir alafenamide and emtricitabine) in rectal tissues | At Day 0, T1 (maximum 3 hours after taking treatment)
  Dosage of the different antiretroviral drugs molecules in rectal tissues

SECONDARY OUTCOMES:
Characterization of the level of the replication (RNA-HIV) in the reservoirs | At Day 0
  Analyze and comparison of the level of viral transcription by measuring the cell-associated HIV- RNA in the different tissues and fluids: lymphoid, rectal, genital secretion, blood and fat biopsies as well as cerebrospinal fluid.
Characterization of the level of infection (DNA-HIV) in the reservoirs | At Day 0
  Analyze and comparison of the reservoir level by measuring the cell-associated total HIV- DNA in the different tissues and fluids
Study of the spatial dynamics of viral quasi-species In the different reservoirs | At Day 0
  Analyze of the spatial dynamics of HIV-DNA and HIV-RNA from Lymphoid, rectal, genital secretion, blood, fat cells by phylogenetic analyses after sequencing Env HIV-DNA and HIV-RNA
Study of the mutations of resistance in the integrase gene | At Day 0
  Description of resistance mutations in Integrase gene which could be linked to suboptimal concentrations of bictegravir
Description for each compartment of the relationship between exposure to therapeutic combinations and the level of infection / viral replication | At Day 0
  Characterization of the relationship between the concentration of bictegravir and backbone drugs with the level of wild type viral replication in the different compartments. Analyze of the impact of backbone drugs associated to bictegravir on viral level production. Correlation between the level of resistant virus replication and the exposure to bictegravir and the backbone drugs. Evaluation by simulation the effect of different dosing regimen of bictegravir (including higher doses) on the level of viral replication and on resistance

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CHERET, Pr, Principal Investigator — Centre de Diagnostic et de Thérapeutique pluridisciplinaire CHU Pointe-à-Pitre/Abymes
Locations (6):
- France (6):
  - Antoine-Beclere Hospita, Clamart
  - Bicetre Hospital, Le Kremlin-Bicêtre
  - Hotel Dieu Hospital, Paris
  - Necker Hospital, Paris
  - Pitie Salpetriere Hospital, Paris
  - Saint Antoine Hospital, Paris